CLINICAL TRIAL: NCT02205892
Title: Clinical Study for the Effectiveness and Safety of Topical Lupeol in Mild to Moderate Acne
Brief Title: Clinical Study for Topical Lupeol in Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dae Hun Suh, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNUH-lupeol
Record Dates: First submitted 2014-07-30; First posted 2014-07-31 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Acne
Keywords: natural product; clinical trial
MeSH Terms: conditions — Acne Vulgaris | interventions — lupeol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lupeol (Active Comparator)
  Interventions: Drug: Lupeol
- Vehicle (Placebo Comparator)
  Interventions: Drug: Placebo vehicle

INTERVENTIONS:
Drug: Lupeol — Patients are supposed to apply 2% lupeol cream to one side of their face two times per day for 4 weeks. Application side is randomly determined.
  Arms: Lupeol
Drug: Placebo vehicle — Patients are supposed to apply their control vehicle cream two times per day to the other side of their face for 4 weeks. Application side is randomly determined.
  Arms: Vehicle

SUMMARY:
Double-blind, randomized,4-week small-scale clinical trial for lupeol in the treatment of inflammatory and non-inflammatory acne lesions in split face fashion

DETAILED DESCRIPTION:
To investigate the clinical efficacy and tolerability of lupeol for the treatment of facial acne, we conducted a small-scale, randomized, double-blinded, split-face clinical trial over the course of 4 weeks. Fifteen of 16 enrolled patients completed the study, in which affected areas on half each patient's face were treated with 2% lupeol twice daily while the other side of the face was treated with a vehicle control. Clinical visits were scheduled at baseline and at 2 and 4 weeks. The primary outcome of the study was the percent change in inflammatory lesions (papules, pustules, and nodules) at 4 weeks. The secondary outcomes were the percent change in non-inflammatory lesions (open and closed comedones) and the change in the Leeds revised acne grading system score at 4 weeks. Adverse events (AEs) were defined as all unintended and harmful signs or symptoms; these were assessed by both patients' self-reporting and physicians' skin examination at each visit. Results were analyzed using intent to treat (ITT) groups. The per-protocol (PP) population consisted of the 15 patients who did not have any major protocol deviations. Last observation carried forward (LOCF) analysis was used to evaluate the primary and secondary outcomes.

** Randomization and blindness process **

At the time of initial presentation, an evaluation of acne severity was performed using both individual counts of inflammatory and non-inflammatory acne lesions and an assessment of the Leeds revised acne grading system score. Then, patients were randomly assigned to either left- or right-sided lupeol application, with the other side of the face assigned to vehicle-control application. A simple random allocation sequence was created using computer-based random number generators with a block size of 4. All dermatologists participating in outcome assessments, a physician assistant managing trial enrollment and administration, medical statisticians analyzing the data, and patients were blinded to the assignments. Randomization codes were strictly secured in a safe in the administration office of the clinical research center until data entry was complete. The integrity of the blinding was ensured by packaging the study- and control products in identical tubes and by requiring a third party (other than the investigator/evaluator) to dispense the medication. In addition, both topical agents were identical in color and odor.

ELIGIBILITY:
Inclusion Criteria:

• Patients over the age 15 years of age or older who were clinically diagnosed with mild to moderate acne vulgaris (Leeds revised acne grading system score 2-7)

Exclusion Criteria:

• Known pregnancy or lactation, any medical illness that might influence the results of the study, a previous history of oral acne medication or surgical procedures including laser treatment within 6 month and topical medication within 4 weeks of study enrollment.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Percent change of inflammatory acne lesion counts | 4 week

SECONDARY OUTCOMES:
Percent change of non-inflammatory acne lesion counts | 4 week

OTHER OUTCOMES:
Change of Leeds revised grade | 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hun Suh, MD, Principal Investigator — Seoul National University Department of Dermatology; Hyuck Hoon Kwon, MD, Study Director — Seoul National University Department of Dermatology; Sun Yong Park, Study Director — Seoul National University Department of Dermatology; Seounguk Min, Study Director — Seoul National University Department of Dermatology; Jae Yoon Jung, Study Director — Seoul National University Department of Dermatology
Locations (1):
- Seoul National University Department of Dermatology, Seoul, South Korea